CLINICAL TRIAL: NCT00775333
Title: Clinical Outcomes of Surgical Release Among Diabetic Patients With Carpal Tunnel Syndrome. A Prospective Study With Matched Controls
Brief Title: Nerve Entrapment in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Niels Thomsen, MD, Dept. of Hand Surgery, Malmo University Hospital, Sweden
Other Study IDs: LU 508-03
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Carpal Tunnel Syndrome; Entrapment Neuropathies; Nerve Compression Syndromes; Diabetes Complications
Keywords: Carpal Tunnel Syndrome; Diabetes; APB strength; Sensory Function; Pillar Pain; Cold Intolerance; Patient Satisfaction
MeSH Terms: conditions — Carpal Tunnel Syndrome; Nerve Compression Syndromes; Diabetes Complications; Diabetes Mellitus; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with diabetes and carpal tunnel syndrome
- 2: Non-diabetic patients with carpal tunnel syndrome
  Interventions: Procedure: Outcome after carpal tunnel release

INTERVENTIONS:
Procedure: Outcome after carpal tunnel release — Follow the outcome after standard carpal tunnel release in diabetic and non-diabetic patients
  Groups: 2

SUMMARY:
The aim of this study is in a prospective, consecutive series of diabetic patients with carpal tunnel syndrome, who are then age and gender matched with non-diabetic patients having idiopathic carpal tunnel syndrome to compare the clinical results after carpal tunnel release.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis was based on clinical history and symptoms of carpal tunnel syndrome
* Confirmed by nerve conduction studies.

Exclusion Criteria:

* Other focal nerve entrapments
* Cervical radiculopathy
* Inflammatory joint disease
* Renal failure
* Thyroid disorders
* Previous wrist fracture
* Long-term exposure to vibrating tools.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a specialized hand clinic
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2003-12; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Sensory function (Semmens-Weinstein), motor function (Abductor Pollicis Brevis (APB)-strength, grip strength) | Baseline, 6 weeks, 12 weeks, 52 weeks

SECONDARY OUTCOMES:
Pillar pain, cold intolerance, and patient satisfaction. | Baseline, 6 weeks, 12 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Dahlin, PHD, Principal Investigator
Locations (1):
- Dept. of Hand Surgery, Malmo University Hospital, Malmo, Sweden